CLINICAL TRIAL: NCT05714943
Title: Web-based Resource for Children and Adolescents About Clinical Research
Brief Title: Website for Adolescents About Pediatric Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovation Research & Training (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Teensinresearch-SBIR-22-002
Record Dates: First submitted 2023-01-24; First posted 2023-02-06 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Healthy; Chronic Illnesses, Multiple
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational website intervention (Experimental): Participants will have access to an intervention between pre-test and post-test assessments. The intervention, DigiKnowIt News: Teen, is an educational website designed to teach youth (12-17 years) about pediatric clinical trials and give parents and youth resources for communication and shared decision-making about research.
  Interventions: Behavioral: DigiKnowIt News: Teen
- Wait-List Control (No Intervention): Participants will not have access to the educational website between the pre-test and post-test assessments. After completing the post-test questionnaires, participants in the wait-list control group will receive access to the intervention (DigiKnowIt News: Teen).

INTERVENTIONS:
Behavioral: DigiKnowIt News: Teen — Participants will interact with a multimedia educational website that will teach them about pediatric clinical trials, including topics such as participant rights and safety and different types of procedures used in trials, and will provide strategies for parent-teen shared decision-making about clinical trials.
  Arms: Educational website intervention

SUMMARY:
The goal of this study is to evaluate the effectiveness of DigiKnowIt News: Teen with parent-adolescent pairs.

DETAILED DESCRIPTION:
Parent-adolescent pairs (N=180) will be recruited to participate in a randomized controlled trial. Parent consent and parent permission and youth assent will be sought. Participant pairs will be randomized into one of two study arms: intervention and wait-list control. All participants will complete a web-based pre-test questionnaire. Youth and parents in the intervention group will then receive access to DigiKnowIt News: Teen for one week. Approximately one week after completing the pre-test questionnaire, all participants will complete a web-based post-test questionnaire (the post-test for the intervention group will include Consumer Satisfaction Questions). Youth and parents in the wait-list control group will then receive access to DigiKnowIt News: Teen for one week. After one week, they will be asked to complete a Consumer Satisfaction Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adult participant is a parent or legal guardian of adolescent participant;
* Adolescent participant is within the ages of 12-17 years;
* Parent-adolescent pair has access to a computer or tablet with internet connection
* Parent-adolescent pair is fluent in English

Exclusion Criteria:

* Adolescent participant has previously participated in a clinical trial after kindergarten.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 255 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Parker, PhD, Principal Investigator — Innovation Research & Training; Tracy Scull, PhD, Principal Investigator — Innovation Research & Training
Locations (1):
- innovation Research & Training, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parker AE, Scull TM, Kennedy KL. Efficacy of DigiKnowItNews: Teen, a multimedia educational website for adolescents about pediatric clinical trials: study protocol for a randomized controlled trial. Trials. 2023 Jun 30;24(1):436. doi: 10.1186/s13063-023-07464-0. PMID 37391773

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 255 enrolled parent-adolescent pairs, 233 met inclusion criteria and were randomized to condition (interview or wait-list control).
Period: Overall Study
Arm/Group | Educational Website Intervention | Wait-List Control
Started | 236 (118 adolescents and 118 parents) | 230 (115 adolescents and 115 parents)
Completed Pretest | 166 (83 adolescents and 83 parents) | 192 (96 adolescents and 96 parents)
Completed | 138 (69 adolescents and 69 parents) | 188 (94 adolescents and 94 parents)
Not Completed | 98 | 42

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Educational Website Intervention | Wait-List Control | Total
Number analyzed (Participants) | 166 | 192 | 358
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The overall sample includes parents and adolescents. The analysis population for adolescent age includes just adolescents and the analysis population for parent age includes just parents.
  years
    Adolescent: number analyzed (Participants) | 83 | 96 | 179
    Adolescent | 14.60 (1.75) | 14.53 (1.52) | 14.56 (1.63)
    Parent: number analyzed (Participants) | 82 | 96 | 178
    Parent | 45.85 (7.04) | 44.08 (6.40) | 44.90 (6.74)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The overall sample includes parents and adolescents. The adolescent sex/gender categories only include adolescents and the parent sex/gender categories only include parents.
  Participants
    Adolescent Male: number analyzed (Participants) | 83 | 96 | 179
    Adolescent Male | 34 | 39 | 73
    Adolescent Female: number analyzed (Participants) | 83 | 96 | 179
    Adolescent Female | 48 | 53 | 101
    Adolescent Non-Binary: number analyzed (Participants) | 83 | 96 | 179
    Adolescent Non-Binary | 1 | 4 | 5
    Parent Male: number analyzed (Participants) | 83 | 96 | 179
    Parent Male | 9 | 9 | 18
    Parent Female: number analyzed (Participants) | 83 | 96 | 179
    Parent Female | 74 | 87 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall sample includes parents and adolescents. The adolescent ethnicity categories include only adolescents and the parent ethnicity categories include only parents.
  Participants
    Adolescent: number analyzed (Participants) | 83 | 96 | 179
    Adolescent: Hispanic or Latino | 21 | 24 | 45
    Adolescent: Not Hispanic or Latino | 62 | 72 | 134
    Adolescent: Unknown or Not Reported | 0 | 0 | 0
    Parent: number analyzed (Participants) | 83 | 96 | 179
    Parent: Hispanic or Latino | 16 | 16 | 32
    Parent: Not Hispanic or Latino | 67 | 80 | 147
    Parent: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall sample includes parents and adolescents. The adolescent race categories include only adolescents and the parent race categories include only parents.
  Participants
    Adolescent: number analyzed (Participants) | 83 | 96 | 179
    Adolescent: American Indian or Alaska Native | 0 | 0 | 0
    Adolescent: Asian | 2 | 2 | 4
    Adolescent: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Adolescent: Black or African American | 9 | 15 | 24
    Adolescent: White | 59 | 65 | 124
    Adolescent: More than one race | 12 | 12 | 24
    Adolescent: Unknown or Not Reported | 1 | 1 | 2
    Parent: number analyzed (Participants) | 83 | 96 | 179
    Parent: American Indian or Alaska Native | 1 | 1 | 2
    Parent: Asian | 4 | 3 | 7
    Parent: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parent: Black or African American | 10 | 15 | 25
    Parent: White | 63 | 72 | 135
    Parent: More than one race | 5 | 5 | 10
    Parent: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 166 | 192 | 358

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Adolescents' Knowledge About Clinical Trials at Week 1
Description: Adolescents will respond to 27 questions that assess their factual knowledge about clinical research (e.g., Which is true of a behavioral treatment trial?). Questions are in multiple choice format (some questions have multiple correct answers), and the total score could range from 0-53 correct. Higher scores indicate more knowledge about clinical research.
Time Frame: Baseline and Week 1
Population: The discrepancy between the overall number of participants analyzed and participant flow is due to imputation. Demographic variables were not imputed so if a participant was missing demographic data, they were not included in the outcome analyses.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 40.32 (.66) | 40.33 (.57)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .99, Regression, Linear

2. Primary Outcome: Change From Baseline in Adolescents' Attitudes About Clinical Trials at Week 1
Description: Adolescents will be asked to respond to 6 questions that assess their positive attitudes about clinical trials (e.g., How do you feel about teens participating in clinical trials?; 1=Not good at all; 2=Not very good; 3=Not sure; 4=Good; 5=Very good). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate more positive attitudes toward clinical trials.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 3.91 (.07) | 3.65 (.05)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .00, Regression, Linear

3. Primary Outcome: Change From Baseline in Adolescents' Beliefs About Clinical Trials at Week 1
Description: Adolescents will be asked to respond to 5 questions about their beliefs about pediatric clinical research (e.g., I believe that clinical trials can help teens; 1=Strongly Disagree; 2=Disagree; 3=Unsure; 4=Agree; 5=Strongly Agree). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate more positive beliefs about clinical trials.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 4.19 (.07) | 4.05 (.05)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .09, Regression, Linear

4. Primary Outcome: Change From Baseline in Adolescents' Self-efficacy to Communicate at Week 1
Description: Adolescents will be asked to respond to 10 questions about their self-efficacy for making decisions about clinical trial participation specific to communicating about clinical trials (e.g., Tell a doctor or researcher if I want to stop the clinical trial; 1 = I cannot do it at all; 5 = I know I can do it.) Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate more self-efficacy about communication.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 4.44 (.07) | 4.39 (.06)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .57, Regression, Linear

5. Primary Outcome: Change From Baseline in Adolescents' Self-efficacy to Gather Information at Week 1
Description: Adolescents will be asked to respond to 9 questions about their self-efficacy for making decisions about clinical trial participation specific to gathering information about clinical trials (e.g., Ask a doctor or researcher questions for more information about clinical trials; 1 = I cannot do it at all; 5 = I know I can do it.) Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate more self-efficacy about gathering information.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 4.15 (.08) | 4.25 (.06)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .32, Regression, Linear

6. Primary Outcome: Change From Baseline in Adolescents' Confidence for Participating in a Clinical Trial at Week 1
Description: Adolescents will be asked to respond to 3 questions about their confidence in participating clinical trials (e.g., I know what rights I have in a clinical trial.; 1=Strongly Disagree; 2=Disagree; 3=Unsure; 4=Agree; 5=Strongly Agree). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate more confidence in participating in clinical trials.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 3.76 (.08) | 3.33 (.07)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .00, Regression, Linear

7. Primary Outcome: Change From Baseline in Adolescents' Procedural Fears at Week 1
Description: Adolescents will be asked to respond to 4 questions related to their perceptions of fear or anxiety about different types of medical procedures, including getting a needle in the arm, injection in the leg, getting a scan, and taking new medicine (1 = Not at all afraid or anxious, 2 = Somewhat afraid or anxious, 3 = Moderately afraid or anxious, 4 = Very afraid or anxious, 5 = Extremely afraid or anxious). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate more fear about procedures.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 2.42 (.09) | 2.42 (.07)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .97, Regression, Linear

8. Primary Outcome: Change From Baseline in Adolescents' Likelihood of Participation at Week 1
Description: Adolescents will be asked to respond to one question about the likelihood of participating in a clinical trial (i.e., If you were asked to be in a clinical trial, how likely would you be to participate?; 1 = Not likely at all; 2 = Not very likely; 3 = Not sure; 4 = Likely; 5 = Very likely). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate greater likelihood of participation in a clinical trial.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 3.64 (.10) | 3.48 (.08)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .21, Regression, Linear

9. Primary Outcome: Change From Baseline in Adolescents' Likelihood of Fear Preventing Participation at Week 1
Description: Adolescents will be asked to respond to one question about the likelihood of their fear preventing them from participating in a clinical trial (i.e., How likely is it that your fearful or anxious feelings could stop you from participating in a clinical trial in the future?; 1 = Not likely; 2 = Somewhat likely; 3 = Moderately likely; 4 = Very likely; 5 = Extremely likely). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate greater likelihood of fear preventing participation in a clinical trial.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 2.71 (.14) | 2.51 (.11)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .27, Regression, Linear

10. Primary Outcome: Change From Baseline in Adolescents' Familiarity With Clinical Trials at Week 1
Description: Adolescents will be asked to respond to one question about their familiarity with clinical trials [How much do you know about pediatric clinical trials (research studies with children under 18; 1 = I don't know anything; 2 = I know a little about them; 3 = I know some things about them; 4 = I know a lot about them; 5 = I know all there is to know about them]. Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate greater familiarity with pediatric clinical trials.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 2.80 (.11) | 2.23 (.09)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .00, Regression, Linear

11. Primary Outcome: Change From Baseline in Adolescents' Willingness to Participate at Week 1
Description: Adolescents will review five research protocols related to a fictitious disease ('meditis') and respond to a question about their willingness to participate in each research study (e.g., If you had meditis, would you agree to enroll in this study?; 1 = Definitely not to 7 = Definitely yes). Responses will be averaged across the five protocols and the minimum scale score is 1 and the maximum scale score is 7. Higher scores indicate greater willingness to participate in the research studies.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 4.45 (.17) | 4.41 (.12)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .86, Regression, Linear

12. Primary Outcome: Change From Baseline in Adolescents' Perceptions of Parent-adolescent Communication Quality at Week 1
Description: Adolescents will be asked to respond to 8 questions related to their perceptions of their relationship quality and communication with their parents (e.g., My parent gives me good advice; 1 = Strongly disagree; 2 = Disagree; 3 = Agree; 4 = Strongly agree). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 4. Higher scores indicate more positive perceptions of relationship quality.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 3.33 (.04) | 3.29 (.04)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .61, Regression, Linear

13. Primary Outcome: Change From Baseline in Parents' Attitudes About Clinical Trials at Week 1
Description: Parents will be asked to respond to 6 questions that assess their positive attitudes about clinical trials (e.g., How do you feel about teens participating in clinical trials?; 1=Not good at all; 2=Not very good; 3=Not sure; 4=Good; 5=Very good). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate more positive attitudes toward clinical trials.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 3.88 (.06) | 3.69 (.05)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .02, Regression, Linear

14. Primary Outcome: Change From Baseline in Parents' Beliefs About Clinical Trials at Week 1
Description: Parents will be asked to respond to 5 questions about their beliefs about pediatric clinical research (e.g., I believe that clinical trials can help teens; 1=Strongly Disagree; 2=Disagree; 3=Unsure; 4=Agree; 5=Strongly Agree). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate more positive beliefs about clinical trials.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 4.18 (.05) | 4.05 (.05)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .08, Regression, Linear

15. Primary Outcome: Change From Baseline in Parents' Likelihood of Participation at Week 1
Description: Parents will be asked to respond to one question about the likelihood of allowing their child to participate in a clinical trial (i.e., If your child were asked to be in a clinical trial, how likely would you be to let them participate?; 1 = Not likely at all; 2 = Not very likely; 3 = Not sure; 4 = Likely; 5 = Very likely). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate greater likelihood of allowing child to participate in a clinical trial.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 3.80 (.09) | 3.61 (.07)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .08, Regression, Linear

16. Primary Outcome: Change From Baseline in Parents' Likelihood of Fear Preventing Participation at Week 1
Description: Parents will be asked to respond to one question about the likelihood of their fear preventing them from allowing their child to participate in a clinical trial (i.e., How likely is it that your fearful or anxious feelings could stop you from allowing your child to participate in a clinical trial in the future?; 1 = Not likely; 2 = Somewhat likely; 3 = Moderately likely; 4 = Very likely; 5 = Extremely likely). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate greater likelihood of fear preventing participation in a clinical trial.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 2.57 (.15) | 2.92 (.11)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .06, Regression, Linear

17. Primary Outcome: Change From Baseline in Parents' Familiarity With Clinical Trials at Week 1
Description: Parents will be asked to respond to one question about their familiarity with clinical trials [How much do you know about pediatric clinical trials (research studies with children under 18; 1 = I don't know anything; 2 = I know a little about them; 3 = I know some things about them; 4 = I know a lot about them; 5 = I know all there is to know about them]. Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate greater familiarity with pediatric clinical trials.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 2.89 (.12) | 2.31 (.09)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .00, Regression, Linear

18. Primary Outcome: Change From Baseline in Parents' Willingness to Participate at Week 1
Description: Parents will review five research protocols related to a fictitious disease ('meditis') and respond to questions about their willingness to let their child participate in each research study (i.e., "If your child had meditis, would you agree to enroll them in this study?"; 1 = Definitely not to 7 = Definitely yes). Responses will be averaged across the five protocols and the minimum scale score is 1 and the maximum scale score is 7. Higher scores indicate greater willingness to allow their child to participate in the research studies.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 4.60 (.10) | 4.62 (.10)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .88, Regression, Linear

19. Primary Outcome: Change From Baseline in Parents' Perceptions of Parent-adolescent Communication Quality at Week 1
Description: Parents will be asked to respond to 16 questions regarding their perceptions of the quality of communication with their adolescent (If my child were in trouble, she/he could tell me; 1 = Strongly Disagree, 2 = Disagree; 3 = Agree; 4 = Strongly Agree). Responses will be averaged and the minimum scale score is 1 and the maximum scale score is 4. Higher scores indicate more positive perceptions of relationship quality.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Educational Website Intervention | Wait-List Control
Number analyzed (Participants) | 82 | 93
units on a scale | 3.15 (.03) | 3.15 (.03)
Statistical Analysis 1: Comparison: Educational Website Intervention vs Wait-List Control; Test type: Superiority; p = .94, Regression, Linear

ADVERSE EVENTS:
Time Frame: From baseline to end of intervention at 1 week
Description: The participants in the study completed web-based questionnaires and utilized an educational website (if in the intervention group). The risks associated with this study were minimal and the participants were not at risk for mortality as a function of participating in this study. Because this study investigated an online behavioral intervention, All-Cause Mortality was not monitored or assessed.
Arm/Group | Educational Website Intervention | Wait-List Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/192
Other Adverse Events (participants affected / at risk) | 0/166 | 0/192

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT05714943/Prot_SAP_000.pdf